CLINICAL TRIAL: NCT02718872
Title: Development and Dissemination of a Tobacco Cessation Training Program for Healthcare Professionals in Spanish-speaking Countries
Brief Title: Tobacco Cessation Training Program in Spanish-speaking Countries
Acronym: FRUITFUL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Català d'Oncologia (Other)
Collaborators: Instituto Oncológico del Oriente Boliviano (Unknown); Instituto de Cancerología y Hospital Dr. Bernardo del Valle (Unknown); Instituto de Enfermedades Respiratoiras INERAM Prof. Dr. Juan Max Boettner (Unknown)
Responsible Party: Principal Investigator, Cristina Martínez Martínez, Doctor, Institut Català d'Oncologia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: FRUITFUL GB-13520139
Record Dates: First submitted 2016-02-02; First posted 2016-03-24 (Estimated); Last update posted 2016-12-22 (Estimated); Status verified 2016-12

CONDITIONS: Smoking; Smoking Cessation
MeSH Terms: conditions — Smoking; Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tobacco cessation online training (Experimental): Six hour smoking cessation online training addressed to health professionals from hospitals in 3 Latin American Countries. Participants are monitored by local coordinators that act as champions. They offer their assistance to log into the online platform, fill out the questionnaires, complete the evaluation, including other technical support. Participants' progress is monitored in real time onto the web platform. The project coordinator at ICO sends a report of the participants progress every other week to coordinators, and if necessary personal emails to motivate students to finish the course and complete the evaluations.
  Interventions: Behavioral: Tobacco cessation online training

INTERVENTIONS:
Behavioral: Tobacco cessation online training — The original course has been developed in the online platform e-oncologia (http://www.e-oncologia.org/en/) based on the in-person courses offered during the last 10 years by the Tobacco Control Unit of the Catalan Institute of Oncology. The theoretical framework underpinning the training program is the Stages of Change Model and the curriculum was developed with the content of numerous meta-analysis and clinical practice guidelines. We created a fully referenced curriculum online, with feedback from an expert advisory group that oriented in the instructional design to ensure the course content was palatable for an online format and aligned with the learning objectives. The final curriculum content of the "Brief Intervention for Smoking Cessation Training Program" is composed of 4 modules.

SUMMARY:
This project is responsive to the identified gap of lack of tobacco cessation training programs in Latin American & Caribbean countries. Currently, smoking rates in the Latin American and Caribbean region are high, and previous surveys show that health professionals do not have enough skills to help smokers to quit. In consequence, in absence of trained health professionals, many smokers who visit health care services are under-treated. The Fruitful Project aims to adapt an original on-line course developed in Spain to the reality of the three Latin American countries (Bolivia, Guatemala and Paraguay) and disseminate evidence-based tobacco cessation interventions among health care professionals.

DETAILED DESCRIPTION:
Tobacco cessation training programs to treat tobacco dependence have measureable effects on patients' smoking. Tobacco consumption in low and middle income countries is increasing, but these countries usually lack measures to face the epidemic, including tobacco cessation training programs addressed to their health professionals and organizations.

Based on a previous online training program for hospital workers in Spain, the Fruitful Study aims are twofold:

1. to adapt the course to the reality of 3 Spanish-speaking low and middle income countries (Bolivia, Guatemala, and Paraguay) and;
2. to evaluate the effectiveness of the program among the participant hospitals and workers.

Investigators use a mixed methods design with a pre-post evaluation (quantitative approach) and in-depth interviews and focus groups (qualitative approach). The main outcomes will be:

1. participants' attitudes, knowledge and behaviors before and after the training and
2. the level of implementation of tobacco control policies within the hospitals before and after the training.

The theoretical framework for this project includes Card's adapting model and Roger's diffusion of innovations model.

This study will show whether it is possible to adapt an online course to the reality of developing countries. In addition, investigator will measure whether an online program will produce changes in tobacco control policies at the organizational level and increase the level of knowledge, attitudes and perception in tobacco cessation at participants' level.

ELIGIBILITY:
Inclusion Criteria:

* Health professionals of the participating centers

Exclusion Criteria:

* No exclusion criteria

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2015-01; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Knowledge, attitudes, and behaviors of trainees | six month
  Trainers' attitudes, knowledge and behaviors will be assessed by using a questionnaire composed of 63-items. The web-site delivered questionnaire is e-mailed to the participants at baseline and 6 months after finishing the training. The questionnaire takes 30-40 minutes to complete. It has been designed according to Sheffer work. The questionnaire gathers information about the provider gender, tobacco use history, previous tobacco cessation education, level of proactivity addressing tobacco use, and perceived success in helping patients stop using tobacco.

SECONDARY OUTCOMES:
Compliance with tobacco control policies in hospitals | one year
  Score in the self-audit questionnaire,

CONTACTS AND LOCATIONS:
Overall Officials: Crisitna Martínez, PhD, Principal Investigator — Institut Català d'Oncologia - Institut d'Investigació Biomèdica de Bellvitge - Universitat de Barcelona ICO-IDIBELL-UB

IPD SHARING:
Plan to Share IPD: No
NO plans for data sharing

REFERENCES:
- [Derived] Martinez C, Company A, Guillen O, Margalef M, Arrien MA, Sanchez C, Caceres de Leon P, Fernandez E; Group of Hospital Coordinators in the Fruitful Project. Adaptation, Implementation Plan, and Evaluation of an Online Tobacco Cessation Training Program for Health Care Professionals in Three Spanish-Speaking Latin American Countries: Protocol of the Fruitful Study. JMIR Res Protoc. 2017 Jan 27;6(1):e7. doi: 10.2196/resprot.6487. PMID 28128731